CLINICAL TRIAL: NCT05789160
Title: Experiential Avoidance as Mechanism of Mindfulness Based Online Intervention in Reducing Emotional Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20220718
Record Dates: First submitted 2023-03-10; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Emotional Distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the MIED group (Experimental): provide standard audio instructions for mindfulness exercises, introduce the nature and law of anxiety, depression and other emotions, the source of anxiety, depression and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression and other emotional problems.
  Interventions: Behavioral: Mindfulness Intervention for Emotional Distress
- the waiting-list group (No Intervention): no treatment.

INTERVENTIONS:
Behavioral: Mindfulness Intervention for Emotional Distress — Mindfulness Intervention for Emotional Distress (MIED) program provide standard audio instructions for mindfulness exercises, introduce the nature and law of anxiety, depression and other emotions, the source of anxiety, depression and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression and other emotional problems.
  Arms: the MIED group

SUMMARY:
This study hopes to explore whether experiential avoidance could be a mediator between mindfulness-based interventions and emotional distress.

DETAILED DESCRIPTION:
The improvement of emotional distress by mindfulness intervention has been supported by a large number of empirical studies. For example, the meta-analysis of the effect of MBSR on people with chronic diseases shows that both anxiety (Hedges' g = 0.47) and depression (Hedges' g = 0.26) in mindfulness intervention group are reduced. Mindfulness-based interventions also have good intervention effect on anxiety (Hedges' g = 0.67) and depression (Hedges' g = 0.48) in the general population. Unfortunately, few studies have used the correct methods to test the mechanism of mindfulness-based interventions in mediation analysis or experiments.

Experiential avoidance refers to the unwillingness to keep in touch with specific personal experiences (such as physical feelings, emotions, thinking, memory, and behavioral tendencies), and to take measures to change the form or frequency of these experiences, as well as the situations that trigger these experiences. Experiential avoidance often has only a short-term effect, but it has no effect in the long run, and may even be unfavorable. The paradox of experiential avoidance is that trying to hide or suppress unpleasant thoughts, feelings and physical feelings will increase the frequency and pain of these same experiences, and will enhance the feeling that they are unreal or out of touch with themselves. In addition, long-term experiential avoidance will interfere with the fun of being completely immersed in any activity, leading to the reduction of the frequency of positive events and the suppression of positive emotions.

Some reviews believe that experiential avoidance is one of the mechanisms of beneficial effects brought by mindfulness. Some cross-sectional studies show that the reduction of empirical avoidance is an important intermediary factor in the path of mindfulness to psychopathology . However, no research has directly tested the mediating role of experiential avoidance in mindfulness-based intervention to alleviate emotional distress, which is also the problem that this study wants to explore. According to Kazdin(2007), in order to prove the timeline principle, that is, the change of experiential avoidance is before the change of emotional distress, we will measure the above variables every week during the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with scores greater than 21 on the Kessler Psychological Distress Scale.

Exclusion Criteria:

* Subjects who could not access the Internet;
* Subjects with insufficient Chinese ability;
* Subjects who have participated in mindfulness based projects for more than 6 weeks before, and / or the current frequency of meditation practice is more than once a week;
* Patients with schizophrenia or psychotic affective disorder, current organic mental disorder, substance abuse disorder and generalized developmental disorder;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Weekly changes of Five Facet Mindfulness Questionnaire during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the 7-week intervention
  The Five Facet Mindfulness Questionnaire is a self-reported questionnaire measuring mindfulness levels. Scores range from 39 to 195, with higher scores indicating higher levels of mindfulness.
Weekly changes of Patient Health Questionnaire during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the 7-week intervention
  The Patient Health Questionnaire is a self-reported questionnaire measuring the degree of being troubled by various common physical symptoms. Scores range from 0 to 30.
  0~4 scores: no physical symptoms; 5~9 scores: mild physical symptoms; 10~14 scores: moderate physical symptoms; 15~30 scores: severe physical symptoms.
Weekly changes of Chinese Perceived Stress Scale during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the 7-week intervention
  The Chinese Perceived Stress Scale is a self-reported questionnaire measuring stress. Scores range from 0 to 56, with higher scores indicating higher levels of stress.
Weekly changes of 10-item Kessler Psychological Distress Scale during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the 7-week intervention
  The 10-item Kessler Psychological Distress Scale is a self-reported questionnaire measuring distress. Scores range from 10 to 50, with higher scores indicating higher levels of distress.
Weekly changes of Overall Anxiety Severity and Impairment Scale during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the 7-week intervention
  The Overall Anxiety Severity and Impairment Scale is a self-reported questionnaire measuring anxiety. Scores range from 0 to 20, with higher scores indicating higher levels of anxiety.
Weekly changes of Overall Depression Severity and Impairment Scale during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the 7-week intervention
  The Overall Depression Severity and Impairment Scale is a self-reported questionnaire measuring depression. Scores range from 0 to 20, with higher scores indicating higher levels of depression.
Weekly changes of Inner Peace Scale during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the 7-week intervention
  The Inner Peace Scale is a self-reported questionnaire measuring peace. Scores range from 0 to 28, with higher scores indicating higher levels of peace.
Weekly changes of Athens Insomnia Scale during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the 7-week intervention
  The Athens Insomnia Scale is a self-reported questionnaire measuring sleepy quality. Scores range from 0 to 24, with lower scores indicating higher levels of sleep quality.

SECONDARY OUTCOMES:
Weekly changes of Brief Experiential Avoidance Questionnaire during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the 7-week intervention
  The Brief Experiential Avoidance Questionnaire is a self-reported questionnaire measuring experiential avoidance. Scores range from 15 to 90, with higher scores indicating higher levels of experiential avoidance.
Weekly changes of Acceptance and Action Questionnaire-II during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the 7-week intervention
  The Acceptance and Action Questionnaire-II is a self-reported questionnaire measuring experiential avoidance. Scores range from 7 to 49, with higher scores indicating higher levels of experiential avoidance.
Weekly changes of the Depression Anxiety Stress Scale during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the 7-week intervention
  The Depression Anxiety Stress Scale is a self-reported questionnaire measuring psychological health. Scores range from 0 to 63, with higher scores indicating lower levels of psychological health.

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Liu, Principal Investigator — Study Principal Investigator
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No